CLINICAL TRIAL: NCT00002883
Title: A PROSPECTIVE RANDOMISED TRIAL OF INDUCTION CHEMOTHERAPY WITH 5-FU CONTINUOUS IV INFUSION AND CISPLATIN VERSUS SURGERY IN RESECTABLE ADENOCARCINOMA OF THE LOW THIRD OF THE ESOPHAGUS AND CARDIOESOPHAGEAL JUNCTION
Brief Title: Surgery With or Without Combination Chemotherapy in Treating Patients With Cancer of the Esophagus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065190; FRE-FNCLCC-94012; EU-96018
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage I gastric cancer; stage II gastric cancer; stage I esophageal cancer; stage II esophageal cancer; adenocarcinoma of the stomach; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Cisplatin; Fluorouracil; Chemotherapy, Adjuvant; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not known whether combining chemotherapy with surgery is more effective than surgery alone.

PURPOSE: Randomized phase III trial to compare the effectiveness of surgery with or without combination chemotherapy in treating patients with cancer of the esophagus.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare survival in patients with operable adenocarcinoma of the lower third of the esophagus or the cardia treated with fluorouracil/cisplatin vs. no chemotherapy prior to surgical resection.
* Assess whether neoadjuvant fluorouracil/cisplatin increases tumor resectability.

OUTLINE: This study is randomized for neoadjuvant chemotherapy. Patients are stratified by performance status, tumor location, and randomizing center.

Patients randomized to no neoadjuvant chemotherapy undergo resection of the tumor with adequate margins and resection of regional lymph nodes (R2 with at least 8 nodal groups recommended).

Patients randomized to neoadjuvant chemotherapy receive fluorouracil and cisplatin at 3-4 week intervals; fluorouracil is given by continuous intravenous infusion for 5 days and cisplatin is given on the first 2 days of fluorouracil administration. Tumor response is assessed after 2 courses; responding patients with no serious toxicity receive a third course. Surgery, as above, is initiated 4-6 weeks after the second or third course of chemotherapy. Upon recovery (within 3-6 weeks), patients who responded to neoadjuvant chemotherapy receive 3-4 additional courses of postoperative chemotherapy (maximum total of 6 courses). Patients whose best response was stable disease are assessed for postoperative radiotherapy.

Patients on either arm with positive resection margins, positive lymph nodes, or equivocal complete resection are referred for postoperative radiotherapy. Further therapy for patients with incomplete resection is at the discretion of the physician.

Patients are followed every 3-4 months for at least 5 years.

PROJECTED ACCRUAL: A total of 250 patients will be entered.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Adenocarcinoma of the lower third of the esophagus or the cardia for which complete resection is feasible

  * Extension to the cardia allowed
  * Cancer of the cardia with extension to the esophagus or stomach allowed

    * No in situ cancer of the cardia
  * No distant metastases

PATIENT CHARACTERISTICS:

Age:

* Not over 75

Performance status:

* WHO 0 or 1

Hematopoietic:

* WBC at least 4,000
* Polymorphonuclear lymphocytes greater than 2,000
* Platelets at least 100,000

Hepatic:

* Not specified

Renal:

* Creatinine less than 1.3 mg/dL (120 micromoles/L)

Cardiovascular:

* No prior myocardial infarction
* No other cardiac contraindication to surgery

Pulmonary:

* No respiratory contraindication to surgery

Other:

* No second malignancy except:
* Basal cell carcinoma of the skin
* Adequately treated in situ carcinoma of the uterine cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for tumors of the cardia

Endocrine therapy

* No prior radiotherapy for tumors of the cardia

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 0 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 1996-10 (Actual); Primary Completion 2006-11 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ychou, MD, PhD, Study Chair — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (1):
- Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier, France

REFERENCES:
- [Result] Boige V, Pignon J, Saint-Aubert B, et al.: Final results of a randomized trial comparing preoperative 5-fluorouracil (F)/cisplatin (P) to surgery alone in adenocarcinoma of stomach and lower esophagus (ASLE): FNLCC ACCORD07-FFCD 9703 trial. [Abstract] J Clin Oncol 25 (Suppl 18): A-4510, 200s, 2007.
- [Result] Ychou M, Pignon JP, Lasser P, et al.: Phase III preliminary results of preoperative fluorouracil (F) and cisplatin (P) versus surgery alone in adenocarcinoma of stomach and lower esophagus (ASLE): FNLCC 94012-FFCD 9703 trial. [Abstract] J Clin Oncol 24 (Suppl 18): A-4026, 2006.